CLINICAL TRIAL: NCT06842862
Title: A Mobile Application to Work on Dysfunctional Beliefs Related to Eating Disorders: a Case Series Study in Three Patients in Remission
Brief Title: Mobile Application for Relapse Prevention in Eating Disorders Beliefs in Three Patients in Remission.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, María Roncero, Associate Professor of Psychology, University of Valencia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2021/162
Record Dates: First submitted 2025-02-18; First posted 2025-02-24 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Eating Disorders
Keywords: Maladaptive beliefs; Relapse prevention; Mobile app; Patients; Case series study
MeSH Terms: conditions — Feeding and Eating Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GGED (Experimental): The patients used the GGED module for 15 days after the first assessment.
  Interventions: Device: GGED

INTERVENTIONS:
Device: GGED — This app is used to work on the dysfunctional beliefs that are associated with eating disorders. The app is made up of a series of levels comprising the topics that are normally worked on in CBT in relation to eating disorders. At each level, affirmations in the form of beliefs appear on the screen, and the person must accept them if they are functional, adaptive and positive; or reject them if they are dysfunctional, maladaptive and negative.

SUMMARY:
This study aims to assess the efficacy of GGED module in preventing relapse in three patients with ED diagnoses in remission. In particular, the objective of the present study is to analyse whether the GGED module diminishes the level of attachment to dysfunctional beliefs related to the maintenance of EDs, which had previously been addressed in CBT therapy. Specifically, an uncontrolled case series design was carried out to assess the changes pre and post use the app. It's expected that after the use of the GGED module for 15 days are, the patients show at the primary level: decrease in the degree of ascription to dysfunctional beliefs associated with ED; and at the secondary level: increase in self-esteem and body satisfaction; decrease in eating symptomatology; and no changes in emotional symptomatology. These results are also expected to be maintained in subsequent follow-ups, at 15 days and a month after to finish the app.

DETAILED DESCRIPTION:
There is a mobile platform, called OCD.app (previously GGtude) which is an evidence-based platform comprising of brief game-like exercises targeting a wide range of psychological symptoms. GGED (GG Eating Disorders) is a module within the app that addresses the core beliefs related to the development and maintenance of eating disorders. In this, a cognitive training exercise is performed: different sentences appear in the form of beliefs, and the person must identify and accept those beliefs that are functional, adaptive and positive, dragging them to the lower part of the screen; and reject those that are dysfunctional, maladaptive and negative dragging them to the upper part of the screen. GGED has shown promising results in reducing maladaptive beliefs in the general adult population and in general adolescent population. In addition, another module that target on obsessive-Compulsive disorder (OCD) has demonstrated its efficacy in preventing relapses in patients diagnosed with OCD in remission. Given that the GGED module has not yet been tested in EDs patients and there is a need for the development of techniques to prevent relapses in these disorders, the objective of the present study is to assess its efficacy in preventing relapse in three patients with ED diagnoses in remission.

ELIGIBILITY:
Inclusion Criteria:

* (1) informed consent signed; (2) a diagnosis of an ED in remission; (3) having received CBT; (4) and access to a mobile device to complete the GGED module.

Exclusion Criteria:

* (1) Not meeting the described inclusion criteria.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2023-09-19 (Actual); Primary Completion 2024-06-24 (Actual); Study Completion 2024-06-24 (Actual)

PRIMARY OUTCOMES:
Change in the degree of ascription to dysfunctional beliefs associated with ED | 15 days and 15 days later
  Score change in eating disorders maladaptive beliefs measured by the Eating Disorder Beliefs Questionnaire (EDBQ). It is composed of 32 items that examines core beliefs about weight, physical appearance and eating that are associated with eating disorders. Items are rated on an analog scale from 0 to 100, being 0 "I do not usually believe this at all" and 100 "I am usually completely convinced that this is true". Higher scores indicate the person has more maladaptive beliefs.
Change in maladaptive body and eating beliefs | 15 days and 15 days later
  Score change in maladaptive body and eating beliefs associated with ED measured by Obsessive Beliefs about Body Size and Eating Survey (OBBSES). It is composed of 57 items, which involve beliefs associated with food, eating, weight and body shape, divided into 5 factors: 1) appearance perfectionism; 2) vulnerability to weight gain; 3) eating control; 4) magical thinking; and, 5) thought control. People have to indicate in each item their degree of agreement in a Likert scale whit 7 point (1= "desagree very much" and 7 = "agree very much"). Higher scores indicate the person has more maladaptive body and eating beliefs.

SECONDARY OUTCOMES:
Change in eating symptomatology | 15 days and 15 days later
  Score change in eating symptoms measured by the Eating Disorder Examination Questionnaire (EDE-Q). It is a 36-item self-report questionnaire with 7-point Likert-type scale ranging from 0 (No day/ No time/ Not at all) to 6 (Every day/ Always/ Completely). It's composed of attitudinal and behavioral items, using for the present study only the attitudinal items (22 items). Higher scores indicate the person has greater presence of eating symptomatology.
Change in body satisfaction | 15 days and 15 days later
  Score change in body satisfaction measured by the Body Appreciation Scale-2 (BAS-2). It is a single-factor questionnaire that evaluates body satisfaction with 10 items on a 5-point Likert scale (1 = Never; 5 = Always). Higher scores indicate the person has more body satisfaction.
Change in self-esteem | 15 days and 15 days later
  Score change in depression symptoms measured by The Patient Health Questionnaire for Depression and Anxiety (PH-4). It consists of 4 items, two for Anxiety and two for Depression, with a 4-point Likert scale (from 0 = "never" to 3 = "almost every day"). Higher scores indicate a greater presence of depression or anxiety symptoms.
Change in depressive and anxious symptomatology | 15 days and 15 days later
  Score change in emotional symptomatology measured by The Depression, Anxiety-Stress Scale (DASS-21). It is composed of 21 items that evaluate emotional negative symptoms: depression, anxiety and stress. It has a Likert scale with 4 points (0 = "Did not apply to me at all" and 3 = "Applied to me very much or most of the time"). In this study only the scale of depression was used, composed of 7 items. Higher scores indicate the person has more emotional symptomatology.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: Yes
Share all IPD that underlie results in a publication.
Time Frame: 3 months after the study is published.
Access Criteria: The variables analyzed will be included in the manuscript in which the RCT data are presented, and will be published on the institutional page of the applicants' university (https://roderic.uv.es/) up to 3 months after the article is published.